CLINICAL TRIAL: NCT04403386
Title: A Prospective Natural History Study of Smoking, Immune Cell Profiles, Epigenetics and COVID-19
Brief Title: Prospective Natural History Study of Smoking, Immune Cell Profiles, Epigenetics and COVID-19
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 200108; 20-E-0108
Record Dates: First submitted 2020-05-23; First posted 2020-05-27 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10-22

CONDITIONS: COVID-19
Keywords: Smoke Exposure; CyTOF Assay; Non-Smoker; Antibody Test; Natural History
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- non-smokers: Participants who have never smoked or do not currently reside with a smoker
- Smokers: Participants who currently smokes and has smoked for at least 5 years

SUMMARY:
Background:

Early evidence in the COVID-19 pandemic suggests that smokers are at a higher risk of having severe effects or dying from the disease. Smoking causes changes in immune cells. Researchers think this may be the reason why smokers are more likely to have severe effects from COVID-19. Researchers want to better understand the interaction between smoking history, the immune system, and COVID-19.

Objective:

To better understand how COVID-19 affects smokers and non-smokers immune systems before and after being infected with the virus.

Eligibility:

Healthy people ages 30-55 who are a smokers or non-smokers who may potentially contract COVID-19

Design:

Participants will be screened over the phone. They will answer questions about their demographics, medical history, medications, and smoking status.

Participants will have up to 6 monthly visits.

At the first visit, participants will have blood tests. Blood will be drawn through a needle in an arm vein. They will provide a saliva sample in a container and have a cheek swab. The participant will also have a nasal swab to see if they currently have COVID-19. Their height and weight will be taken. They will complete questionnaires about their medical history and smoking status.

Participants will then have monthly visits. They will have blood draws to test for COVID-19 antibodies. They will provide a saliva sample in a container and have a cheek swab. The participant will also have a nasal swab to see if they currently have COVID-19.

These visits will occur 4 times or until they have a positive antibody result.

Participants will have a final visit. They will have blood tests. They will provide a saliva sample in a container and have a cheek swab. The participant will also have a nasal swab to see if they currently have COVID-19.

If at any time participants test positive for a COVID-19, they will be rescheduled 14 days or more after they no longer have symptoms....

DETAILED DESCRIPTION:
Study Description:

This study is a prospective, longitudinal, observational, single-center, exploratory study to collect samples and data that will enable explorations of the interaction between smoking, immune system characteristics and Coronavirus Disease 2019 (COVID-19). This study will collect baseline samples and data prior to COVID-19 infection required to explore these interactions prospectively.

Early evidence in the COVID-19 pandemic suggests that smokers have higher risk for morbidity and mortality associated with COVID-19 infection. We have identified smoking-associated altered epigenetics, transcription and changes in immune cell profiles.

Smoking exposure drives loss of naive CD8+ T cells and increases in senescent CD8+ T cells and these effects are signs of immune system dysfunction. We propose that the immune system senescence associated with prior smoking is a susceptibility factor in COVID-19 morbidity.

Objectives:

Primary Objective:

To prospectively collect biospecimens and data at baseline and longitudinally in an identified fashion from eligible participants and retain for future use to better understand the interaction between smoking history, immune cell profiles and the natural history of COVID-19 morbidity. We hypothesize that senescent CD8 T cells will be higher in smokers who develop COVID-19.

To test this hypothesis, we will establish a bank of cryopreserved peripheral blood mononuclear cells (PBMCs) from before and after COVID-19 exposure from smokers and nonsmokers and use mass cytometry (CyTOF) to analyze detailed immune profiles, test if the frequency of senescent CD8 T cells is higher among smokers who develop COVID-19 (antibody positivity) relative to those who do not develop COVID-19 positivity.

Exploratory Objective:

To compare potential immunological biomarkers of susceptibility to viral infection with genetic, epigenetic and other biological characteristics measured in blood before, at one timepoint after recovery from COVID-19 illness and/or post-COVID-19 vaccination and develop assays that indicate immune cell dysfunction and COVID-19 susceptibility.

Endpoints:

Primary Endpoint:

Levels of senescent CD16+CD8+ T cells before COVID-19 and time to COVID-19 morbidity.

Exploratory Endpoints:

1. Smoking exposure biomarkers
2. Immune cell profiles identified by CyTOF assays or other single cell assays
3. Transcriptional profiles from immune cell subtypes
4. DNA methylation profiles of candidate genes in immune cell subtypes

Study Population:

Male and female participants aged 30 to 55 years old, generally healthy with a history of smoking (n=60) and nonsmoking (n=30).

Description of Sites/Facilities Enrolling Participants:

All visits will be conducted at the NIEHS Clinical Research Unit (CRU) in Durham, North Carolina, USA.

Study Duration: Estimated time from enrollment to completion of data analyses is 24 months.

Participant Duration:

Estimated average amount of time for a participant to complete all study visits is 6 months.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Stated willingness to comply with all study procedures and availability for the duration of the study
2. Male and females
3. Age 30 to 55 years
4. Able to travel to study visits at the NIEHS CRU for required study visits
5. Body mass index (BMI) range between 18 and 35 at enrollment
6. Must self-identify as a current smoker (cigarettes and/or use of an e-cigarette/vaping device), have smoked for 5 years or longer or identify as a non-smoker, having never used of any other forms of tobacco, nicotine, or smoked marijuana and not currently residing with a smoker (There may be circumstances where the investigator will still want to include the par icipant (for example when a participant has smoked a couple times in the past and the Investigator feels it has been long enough that they can be included as a nonsmoker or they smoked for over 5 years and quit for a day so they can still be included as a smoker). However, these are expected to be rare and will need to be assessed on a case by case basis by the Investigator to maintain scientific integrity)

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. History of confirmed COVID-19 infection
2. Current diagnosis of cancer or prior history of cancer, with the exception of nonmelanoma skin cancer because nonmelanoma skin cancers are not relate to tobacco smoking and are very common (approximately 20% of US population will develop these). Treatments are generally topical creams or minor surgery with a very high cure rate. If these treatments occurred in the past, they are unlikely to impact the outcomes we are measuring in our pre and post disease study design
3. Bleeding disorder or any reason that a blood sample cannot be provided
4. Current pregnancy or lactation, by participant verbal confirmation.
5. Any condition that, in the investigator's opinion, places the participant at undue risk for complications associated with required study procedures

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Healthy smokers and nonsmokers age 30-55 years
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
Levels of senescent CD16+CD8+ T cells prior to COVID-19 disease and time to COVID-19 disease morbidity (antibody positvity). | At pre and post COVID 19 infection
  The presence of elevated senescent CD16+CD8+ T cells is an indication of immune dysfunction and could be a susceptibility factor.

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Garantziotis, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- NIEHS Clinical Research Unit (CRU), Research Triangle Park, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided
Undecided: It is not yet known if there will be a plan to make IPD available

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-E-0108.html

DOCUMENTS (1):
  • Informed Consent Form (2022-07-26): https://cdn.clinicaltrials.gov/large-docs/86/NCT04403386/ICF_000.pdf